CLINICAL TRIAL: NCT02047838
Title: Impact on Ovarian Reserve of Second Laparoscopic Surgery for Recurrent Unilateral Endometriomas: a Case-control Study.
Brief Title: Second Laparoscopic Surgery for Recurrent Unilateral Endometriomas.
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Umberto Leone Roberti Maggiore, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: Lillo 01/2014
Record Dates: First submitted 2014-01-25; First posted 2014-01-28 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Endometrioma; Endometriosis; Surgery
MeSH Terms: conditions — Endometriosis | interventions — Anti-Mullerian Hormone; Follicle Stimulating Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases.: Patients with recurrent unilateral endometrioma who were previously operated for the same condition.
  Interventions: Other: Anti-mullerian hormone (AMH) level dosage.; Other: Follicle-stimulating hormone (FSH) level dosage.; Other: Antral follicle count (AFC).
- Controls.: Patients previously operated for unilateral endometrioma without recurrence.
  Interventions: Other: Anti-mullerian hormone (AMH) level dosage.; Other: Follicle-stimulating hormone (FSH) level dosage.; Other: Antral follicle count (AFC).

INTERVENTIONS:
Other: Anti-mullerian hormone (AMH) level dosage.
Other: Follicle-stimulating hormone (FSH) level dosage.
Other: Antral follicle count (AFC).

SUMMARY:
This retrospective case-control study was performed in an Academic centre for the diagnosis and treatment of endometriosis. It included patients with recurrent unilateral endometriomas who were previously operated for the same condition (cases) and patients without recurrency who previously underwent surgery for unilateral endometrioma (controls). The primary outcome of the study was to assess the impact on ovarian reserve of second surgery for recurrent unilateral endometriomas. The evaluation of ovarian reserve was performed by assessing serum anti-mullerian hormone (AMH) level, serum follicle-stimulating hormone (FSH) level, 17-beta estradiol level and antral follicle count (AFC).

ELIGIBILITY:
Inclusion Criteria:

* reproductive age (at the time of both surgical procedures);
* two surgical procedures on the same ovary (stripping of endometrioma with
* largest diameter ≥ 4 cm; cases) performed at our Institution;
* one surgical procedures (stripping of endometrioma with largest diameter ≥ 4 cm; controls) performed at our Institution;
* histological diagnosis of ovarian endometriomas;
* complete assessment of ovarian reserve at routinary follow-up at our institution.

Exclusion Criteria:

* patients aged ≥ 40 years at the time of primary surgery;
* surgical procedures on the contralateral ovary (at primary or second-line surgery);
* previous salpingectomy or hysterectomy;
* unilateral ovariectomy at the time of first or second surgery;
* ultrasonographic diagnosis of persistent endometrioma after first surgery;
* additional surgical procedures for endometriomas or for other ovarian diseases before first surgery and between first and second surgery;
* hormonal treatment within 3 months from ovarian reserve assessment;
* patients followed-up < 3 months after second-line surgery (for cases).
* pregnancy and/or breastfeeding during the study period.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: In this study were recruited women referred to an academic centre for the diagnosis and treatment of endometriosis.
  Cases were patients undergoing second surgery for recurrent unilateral endometrioma.
  Controls were patients previously operated for unilateral endometrioma.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Anti-mullerian hormone (AMH) level. | In cases, anti-mullerian hormone (AMH) level was determined 3 months after second laparoscopic surgery. In controls, AMH levels was determined in the the fertility assessment performed during follow-up (matched to the correspondent case).

SECONDARY OUTCOMES:
Follicle-stimulating hormone (FSH) level. | In cases, follicle-stimulating hormone (FSH) level was determined 3 months after second laparoscopic surgery. In controls, FSH levels was determined in the the fertility assessment performed during follow-up (matched to the correspondent case).
17-beta estradiol level. | In cases, 17-beta estradiol level was determined 3 months after second laparoscopic surgery. In controls, 17-beta estradiol level was determined in the the fertility assessment performed during follow-up (matched to the correspondent case).
Antral follicle count (AFC). | In cases, antral follicle count (AFC) was determined 3 months after second laparoscopic surgery. In controls, antral follicle count was determined in the the fertility assessment performed during follow-up (matched to the correspondent case).

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, PhD, Study Director — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy; Umberto Leone Roberti Maggiore, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Ligury, Italy

REFERENCES:
- [Derived] Ferrero S, Scala C, Racca A, Calanni L, Remorgida V, Venturini PL, Leone Roberti Maggiore U. Second surgery for recurrent unilateral endometriomas and impact on ovarian reserve: a case-control study. Fertil Steril. 2015 May;103(5):1236-43. doi: 10.1016/j.fertnstert.2015.01.032. Epub 2015 Feb 11. PMID 25681854